CLINICAL TRIAL: NCT00684255
Title: Reduced Intensity Conditioning And Allogeneic Stem Cell Transplantation in Patients With Medically Refractory Systemic Lupus Erythematosus and Medically Refractory Systemic Sclerosis (SSc)
Brief Title: Reduced Intensity Transplant in Medically Refractory Systemic Lupus Erythematosus (SLE) and Systemic Sclerosis (SSc)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: inactive
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAB1324; CHNY-01-511 (Other: CU)
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2009-12-02 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-02

CONDITIONS: Systemic Lupus Erythematosus; Systemic Sclerosis
Keywords: Autoimmune Disease; Reduced Intensity Transplant
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Autoimmune Diseases | interventions — fludarabine; Busulfan; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduced Intensity Regimen for Refractory SLE (Experimental): RI regimen of fludarabine/busulfan and Alemtuzumab (FBA) followed by AlloSCT in selected patients with medically refractory Systemic Lupus Erythematosus (SLE).
  Interventions: Procedure: Reduced Intensity Allogeneic Transplant; Drug: Fludarabine; Drug: Busulfan; Drug: Campath
- Reduced Intensity Regimen for SSc (Experimental): RI regimen of fludarabine/busulfan and Alemtuzumab (FBA) followed by AlloSCT in selected patients with Systemic Sclerosis (SSc).
  Interventions: Procedure: Reduced Intensity Allogeneic Transplant; Drug: Fludarabine; Drug: Busulfan; Drug: Campath

INTERVENTIONS:
Procedure: Reduced Intensity Allogeneic Transplant — Eeduced intensity allogeneic stem cell transplantation with a fludarabine/busulfan/alemtuzumab conditioning regimen is anticipated to result in mixed and/or complete donor chimerism and potentially alter the natural history and outcome of patients with medically refractory Systemic Lupus Erythematosus (SLE) or Systemic Sclerosis (SSc).
Drug: Fludarabine — Fludarabine 30 mg/m2 Day -7, -6, -5, -4, -3, -2
Drug: Busulfan — Busulfan 3.2 mg/kg Days _8, -7, -6, -5
Drug: Campath — Campath: 2 mg/m2 Day -5; 6 mg/m2 Day -4, -3; 20 mg/m2 Day -2
  Other Names: Alemtuzumab

SUMMARY:
The purpose of this study is to determine if a reduced intensity (RI) (non-myeloablative) chemoimmunotherapy followed by Allogeneic Stem Cell Transplantation AlloSCT (matched family donors and matched unrelated cord blood donors) will be well tolerated.

DETAILED DESCRIPTION:
This is to test whether a reduced intensity will result in a high degree of mixed or complete donor chimerism and stabilization of autoimmune disease in a select group of patients with medically refractory SLE or SSc.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse Systemic Sclerosis and variants as per ACR criteria
* Medically refractory disease
* Adequate Organ Function - Pulmonary function
* Renal function, Cardiac function defined as:
* SGOT (AST) or SGPT (ALT) <5 x upper limit of normal
* Diagnosis of SLE - Medically refractory disease

Exclusion Criteria:

* Karnofsky/Lansky <60%

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- See also: (Click on "Morgan Stanley Children's Hospital" and then "Clinical Services" and then "Blood & Marrow Transplantation") — http://www.childrensnyp.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study closed due to low accrual.
Groups:
- Reduced Intensity Regimen SSc: Reduced Intensity Regimen Medically Refractory Systemic Sclerosis (SSc)
Period: Overall Study
Arm/Group | Reduced Intensity Regimen SSc
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Systemic Sclerosis (SSc): Reduced Intensity Regimen Medically Refractory Systemic Sclerosis (SSc)
Arm/Group | Systemic Sclerosis (SSc)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants] — Subjects 7-17yrs will be enrolled
  Participants
    <=18 years | 1
    Between 18 and 65 years | 0
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Toxicity
Description: Toxicity associated with reduced intensity regimen of fludarabine/busulfan and Campath followed by allogeneic stem cell transplant in patients with medically refractory Systemic Lupus Erythematosus (SLE) or SSc is measured.
Time Frame: 1 year
Groups:
- Medically Refractory Systemic Lupus Erythematosus (SLE): Reduced Intensity Regimen of Fludarabine/Busulfan and Campath Followed by alloSCT in patients with Medically Refractory Systemic Lupus Erythematosus (SLE)
- Systemic Sclerosis (SSc): Reduced Intensity Regimen of Fludarabine/Busulfan and Campath Followed by alloSCT in patients with Systemic Sclerosis (SSc)
Arm/Group | Medically Refractory Systemic Lupus Erythematosus (SLE) | Systemic Sclerosis (SSc)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Chimerism
Description: Percentage(%) of mixed and/or complete donor chimerism has been measured at different time points.
Time Frame: 1 year
Reporting Status: Not Posted
Measure: Number (Standard Deviation); unit: participants

3. Secondary Outcome: Immune Reconstitution.
Description: Peripheral blood for immune reconstitution for T-cell, B-cell and NK cells to be obtained for measurement of cell.
Time Frame: 1 year
Reporting Status: Not Posted
Measure: Number (Standard Deviation); unit: participants

4. Secondary Outcome: Progression Free and Overall Survival.
Description: Probability of progression free and overall survival will be measured.
Time Frame: 1 year
Reporting Status: Not Posted
Measure: Number (Standard Deviation); unit: participants

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Reduced Intensity Regimen SSc
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Study closed due to low accrual. Did not meet enrollment goals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No